CLINICAL TRIAL: NCT05820711
Title: A Phase I Dose-Escalation Trial of Mesenchymal Stromal Cells in Patients With Xerostomia After Radiation Therapy for Head and Neck Cancer
Brief Title: Study Transplanting Bone Marrow Cells Into Salivary Glands to Treat Dry Mouth Caused by Radiation Therapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0194; UW21144 (Other: UW Madison); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); Protocol Version 9/13/2024 (Other: UW Madison); 4UH3DE030431-02 (NIH); A533300 (Other: UW Madison)
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer; Xerostomia
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stem Cell (MSC) injection (Experimental)
  Interventions: Drug: MSC

INTERVENTIONS:
Drug: MSC — Injection of MSCs into submandibular glands at pre-specified dose level:
  * Dose -1: 5 (4 - 6) x10^6 MSCs (to be used only if Dose level 1 is not tolerated) per gland (0.5 ml)
  * Dose 0: 10 (8 - 12) x10^6 MSCs per gland (1 ml)
  * Dose 1: 20 (16 - 24) x10^6 MSCs per gland (2 ml)

SUMMARY:
The goal of this clinical research study is to evaluate the safety and tolerability of injecting certain cells that you produce in your bone marrow called mesenchymal stem cells (MSCs) into your salivary glands.

Participants will have head and neck cancer that was treated with radiation therapy, and in this study will:

* Undergo a collection of bone marrow using a needle;
* Donate saliva;
* Undergo a salivary gland ultrasound; and,
* Complete questionnaires that ask about dry mouth

Participants can expect to be in this study for up to 30 months.

There is no expanded access program available per this protocol.

ELIGIBILITY:
Inclusion Criteria:

* History of histological diagnosis of head and neck cancer (HNC) that was treated with radiation therapy and currently clinically or radiologically no evidence of disease (NED)
* Xerostomia, defined as patient reported salivary function (pre-treatment) ≤ 80% of healthy (pre-radiation)
* ≥ 18 years of age, ≤ 90 years of age.
* Patients ≥ 2 years from completion of radiation therapy for HNC
* Karnofsky performance status ≥ 70, patient eligible for bone marrow aspirate with wakeful anesthesia
* Willing and able to give informed consent
* Radiographically confirmed submandibular gland(s)

Exclusion Criteria:

* Salivary gland disease (i.e., sialolithiasis)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability: Determination of Recommended Phase 2 Dose (RP2D) | Up to 1 month post-injection
  RP2D (also called the maximum tolerated dose) of MSCs determined by the proportion of subjects experiencing dose limiting toxicity (DLT)
Safety and Tolerability: Number of subjects with pain >5 on a 0-10 point scale | 1 month post-injection
  Incidence of pain assessed as greater than 5 on standard 0-10 point pain scale (0=not at all to 10=worst pain imaginable)
Safety and Tolerability: Number of Serious Adverse Events | Up to 1 month post-injection
  Incidence of any serious adverse event
Safety and Tolerability: Number of Treatment-Emergent Pre-Specified Adverse Events | Up to 1 month post-injection
  Incidence of pre-specified adverse events

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline to 24 months post-injection
  Efficacy of MSC assessed through University of Michigan Xerostomia Related Quality of Life (XeQOL) scale, which is a 15-item assessment scale with 4 domains. The score is the average of all responses of all domains and can range from 0 to 4, where higher scores indicate increased xerostomia burden.
Change in Quality of Life | Baseline to 24 months post-injection
  Efficacy of MSC assessed through the MD Anderson Dysphagia Index (MDADI), which is a 20-item questionnaire designed for evaluating the impact of dysphagia (swallowing ability). Scores range from 20 (extremely low functioning) to 100 (high functioning).
Change in Quality of Life | Baseline to 24 months post-injection
  Efficacy of MSC assessed through VAS xerostomia questionnaire, which is an 8-item questionnaire that measures the perception of dry mouth. Scores range from 0-10, with 0 being low dryness and 10 being high dryness.
Change in salivary production | Baseline to 24 months post-injection
  Saliva production will be measured by having participants chew inert gum base to the pace of a metronome (70 beats per minute) while expectorating saliva (without swallowing) into the saliva collection aid for 5 minutes total40. Cryovials will be weighed before and after collection and the difference in weight (g) will represent the amount of saliva produced in 5 minutes for each condition.
Shear wave velocity with acoustic radiation force impulse | 3, 6, and 12 months post-injection
  Assess imaging characteristics of submandibular glands after MSC, measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Randall Kimple, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Jacques Galipeau, MD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States